CLINICAL TRIAL: NCT02547558
Title: Pulmonary Gas Exchange Response to Indacaterol in Stable Symptomatic Chronic Obstructive Pulmonary Disease Patients
Brief Title: Pulmonary Gas Exchange Response to Indacaterol in COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Isabel Blanco, MD, PhD, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IndaEPOC
Record Dates: First submitted 2015-09-04; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Indacaterol; Pulmonary gas exchange; Long-acting bronchodilators
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Blood Gas Analysis; Hydrogen-Ion Concentration; Cardiac Output; Respiratory Rate; Heart Rate; Blood Pressure; Oxygen; Carbon Dioxide; indacaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indacaterol (Experimental): Drug:
  -Indacaterol, inhaled, single dose, 300 mcg
  Diagnostic Interventions:
  * Arterial blood gases
  * Cardiac output
  * Vital signs
  * Exhaled breath
  * Spirometry
  Interventions: Procedure: Arterial blood gases; Procedure: Cardiac Output; Procedure: Vital signs; Procedure: Exhaled breath; Procedure: Spirometry; Drug: Indacaterol

INTERVENTIONS:
Procedure: Arterial blood gases — Measured through radial arterial catheter
  Other Names: PaO2; PaCO2; pH; AaPO2
Procedure: Cardiac Output — Measured through bioimpedance: FloTrac pressure transducer (FloTrac sensor; Edwards Lifesciences) using the third-generation (3.01) FloTrac software for continuous CO display.
  Other Names: CO
Procedure: Vital signs — As measured in clinical practice
  Other Names: Respiratory rate; Heart rate (HR); Systemic arterial pressure
Procedure: Exhaled breath — Were recorded using a pneumotachograph (CPX/D; Med Graphics, St. Paul, MN, U.S.A.).
  Other Names: Oxygen; Carbon dioxide
Procedure: Spirometry — In a daily calibrated spirometer.
  Other Names: FEV1; VFC
Drug: Indacaterol — Indacaterol Breezhaler@ 300 mcg (1 inhalation)
  Other Names: Ultra long acting beta 2 agonist

SUMMARY:
To evaluate the pulmonary gas exchange response to a therapeutic high dose of inhaled indacaterol (300 mcg) in 20 outpatients with stable symptomatic COPD B and D GOLD 2011 groups.

Measurements on a single day before and after 60 and 120 minutes of indacaterol will include arterial PO2, PaCO2 and pH. AaPO2; SaO2 (by pulse oximetry) and oxygen and carbon dioxide in exhaled breath, systemic arterial pressure and heart rate will also be measured/calculated. Cardiac output will be directly measured by bio-impedance.

DETAILED DESCRIPTION:
The investigators hypothesize that in stable chronic obstructive pulmonary disease (COPD) patients the interaction between intrapulmonary and extrapulmonary determinants contributing to gas exchange abnormalities after indacaterol will ultimately preserve arterial oxygenation (primary end-point outcome).

The study will include 20 outpatients with diagnosis of stable COPD in GOLD 2011 groups B and D (10 each), without frequent exacerbations (≥2 in the previous year). Patients with a COPD exacerbation within 3 months of study, use of long-term oxygen therapy and associated conditions or serious comorbidities (i.e., asthma, bronchiectasis, lung cancer and/or cardiovascular diseases) will be excluded.

Each patient will be studied on a single day. All subjects will remain on their regular treatment for the study. Subjects will be required to withhold SABAs for at least 12 h and LABAs and theophylline for at least 24 h before study. During measurements, patients will breath room air and will be seated in an armchair. Measurements will be performed before and 60 and 120 min after a single dose administration of indacaterol Breezhaler@ 300 mcg (1 inhalation).

After ensuring steady-state conditions, as assessed by stability (± 5%) of both ventilatory and hemodynamic variables, and by the close agreement (within ± 5%) between duplicate of mixed expired and arterial oxygen and carbon dioxide, a set of duplicate measurements for each variable will be obtained at each time point.

Blood samples will be collected through a catheter inserted under local anesthesia into the radial artery. Samples of blood (5 ml) will be removed for measurement of arterial O2 tension (PaO2), CO2 tension (PaCO2) and pH; alveolar-arterial PO2 difference (A-a)DO2, oxygen saturation (SaO2), and VO2, VCO2, Ve, respiratory rate (f), systemic arterial pressure (Psa), and heart rate (HR) will be measured or calculated, as previously described.

Cardiac output will be directly measured by bio-impedance. Spirometry values will be recorded from the history records of each patient. All measurements will be performed in the Centre de Diagnòstic Respiratori (CDR), Servei de Pneumologia, Institut del Tòrax, Hospital Clínic, Barcelona.

The primary outcome will be the PaO2 change after indacaterol at each analysis time. Based on a previous study in stable severe COPD patients using nebulized salbutamol during convalescence of exacerbation, Polverino et al. calculated that for a significant PaO2 fall of the order of 8 mmHg, a sample of 6 subjects is needed; this number was increased to 20 patients to ensure better data.

Secondary outcomes were changes in PaCO2, pH, the calculated D(A-a)DO2 and the response of cardiac output.

Results will be expressed as mean (±SEM) or median (95% CI). The effects of indacaterol on each of the end-point variables will be assessed by one-way repeated measures analysis of variance (ANOVA). Paired t tests and Pearson's correlation tests will be used as appropriate. All significances will be set at p<0.05, without correction for multiple tests.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with COPD diagnosis according to GOLD 2011 criteria (VEF1/CVF less than 70%), groups B and D.

Exclusion Criteria:

* Conditions or serious comorbidities (i.e., asthma, bronchiectasis, lung cancer and/or cardiovascular diseases).
* Patients with frequent exacerbations (2 or more exacerbations in the past year).
* History of acute COPD exacerbation in the previous 3 months.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Change in PaO2 after indacaterol. | 60 and 120 minutes

SECONDARY OUTCOMES:
Change in PaCO2 after indacaterol. | 60 and 120 minutes
Change in D(A-a)DO2 after indacaterol. | 60 and 120 minutes
Change in pH after indacaterol. | 60 and 120 minutes
Change in cardiac output after indacaterol. | 60 and 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Blanco, MD, PhD, Principal Investigator — Hospital Clínic
Locations (1):
- Hospital Clínic, Barcelona, Spain

REFERENCES:
- [Background] Viegas CA, Ferrer A, Montserrat JM, Barbera JA, Roca J, Rodriguez-Roisin R. Ventilation-perfusion response after fenoterol in hypoxemic patients with stable COPD. Chest. 1996 Jul;110(1):71-7. doi: 10.1378/chest.110.1.71. PMID 8681669
- [Background] Pillet O, Manier G, Castaing Y. Anticholinergic versus beta 2-agonist on gas exchange in COPD: a comparative study in 15 patients. Monaldi Arch Chest Dis. 1998 Feb;53(1):3-8. PMID 9632900
- [Background] Whale CI, Sovani MP, Mortimer K, Oborne J, Cooper S, Harrison TW, Tattersfield AE. Effects of rac-albuterol on arterial blood gases in patients with stable hypercapnic chronic obstructive pulmonary disease. Br J Clin Pharmacol. 2006 Aug;62(2):153-7. doi: 10.1111/j.1365-2125.2006.02604.x. PMID 16842389
- [Background] Kew KM, Mavergames C, Walters JA. Long-acting beta2-agonists for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2013 Oct 15;2013(10):CD010177. doi: 10.1002/14651858.CD010177.pub2. PMID 24127118
- [Background] Kew KM, Dias S, Cates CJ. Long-acting inhaled therapy (beta-agonists, anticholinergics and steroids) for COPD: a network meta-analysis. Cochrane Database Syst Rev. 2014 Mar 26;2014(3):CD010844. doi: 10.1002/14651858.CD010844.pub2. PMID 24671923
- [Background] Khoukaz G, Gross NJ. Effects of salmeterol on arterial blood gases in patients with stable chronic obstructive pulmonary disease. Comparison with albuterol and ipratropium. Am J Respir Crit Care Med. 1999 Sep;160(3):1028-30. doi: 10.1164/ajrccm.160.3.9812117. PMID 10471636
- [Background] Zafar MA, Droege C, Foertsch M, Panos RJ. Update on ultra-long-acting beta agonists in chronic obstructive pulmonary disease. Expert Opin Investig Drugs. 2014 Dec;23(12):1687-701. doi: 10.1517/13543784.2014.942730. Epub 2014 Aug 19. PMID 25139313
- [Background] Roskell NS, Anzueto A, Hamilton A, Disse B, Becker K. Once-daily long-acting beta-agonists for chronic obstructive pulmonary disease: an indirect comparison of olodaterol and indacaterol. Int J Chron Obstruct Pulmon Dis. 2014 Jul 31;9:813-24. doi: 10.2147/COPD.S59673. eCollection 2014. PMID 25114521
- [Background] Cazzola M, Segreti A, Stirpe E, Puxeddu E, Ora J, Rogliani P, Matera MG. Effect of an additional dose of indacaterol in COPD patients under regular treatment with indacaterol. Respir Med. 2013 Jan;107(1):107-11. doi: 10.1016/j.rmed.2012.09.022. Epub 2012 Oct 18. PMID 23083839
- [Background] Gabrijelcic J, Casas A, Rabinovich RA, Roca J, Barbera JA, Chung KF, Rodriguez-Roisin R. Formoterol protects against platelet-activating factor-induced effects in asthma. Eur Respir J. 2004 Jan;23(1):71-5. doi: 10.1183/09031936.03.00057803. PMID 14738234
- [Background] Polverino E, Gomez FP, Manrique H, Soler N, Roca J, Barbera JA, Rodriguez-Roisin R. Gas exchange response to short-acting beta2-agonists in chronic obstructive pulmonary disease severe exacerbations. Am J Respir Crit Care Med. 2007 Aug 15;176(4):350-5. doi: 10.1164/rccm.200612-1864OC. Epub 2007 Apr 12. PMID 17431221